CLINICAL TRIAL: NCT00961090
Title: A Phase 2 Study of Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Primary Glial Neoplasms of the Brain.
Brief Title: Safety Study of Aminolevulinic Acid (ALA) to Improve Visibility of Brain Tumors During Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew R Quigley (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Matthew R Quigley, administrator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104974
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2015-09

CONDITIONS: Glioblastoma
Keywords: Brain tumor; glioma; surgical resection; ALA; ultraviolet light
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-Arm (Other): Single-Arm All subjects received 20mg/kg of Aminolevulinic Acid diluted in 50cc of water, orally, approximately 3 hours prior to surgery.
  Interventions: Drug: Aminolevulinic Acid

INTERVENTIONS:
Drug: Aminolevulinic Acid — 20 mg/kg mixed in 50cc water and taken orally 3 hours prior to surgery
  Other Names: ALA

SUMMARY:
A one time oral dose of ALA is taken before surgery. The medication makes the tumor visible under ultraviolet light which allow the surgeon to see more of the tumor for a more complete removal.

DETAILED DESCRIPTION:
Patients with primary neoplastic brain tumors (Grades II-IV) will participate in this trial. Each patient will have been evaluated and found to have such a tumor by history and recent imaging studies (MRI) and deemed a surgical candidate based on current neurosurgical standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Suspected primary brain tumor
* 18 years of age or more
* Normal marrow and organ function
* Eastern Cooperative Group performance status ≤ 2
* Women of childbearing potential must use adequate birth control
* Ability to understand and willingness to sign a written informed consent form
* Life expectancy not a consideration

Exclusion Criteria:

* Receiving any other investigational agents
* History of allergic reactions to ALA
* Personal or family history of porphyrias
* Liver disease in the past year
* Uncontrolled intercurrent illness
* Pregnant or lactating women
* Inability to undergo MRI with contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-09; Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-23 (Actual)

PRIMARY OUTCOMES:
More complete resection of malignant brain tumors | 3-7 days

SECONDARY OUTCOMES:
Safety of drug | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Quigley, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States